CLINICAL TRIAL: NCT05980013
Title: Evaluation of Physiological Variables and Detection of Blood Loss in Healthy Adults With Different Subject Positioning by the Zynex Cardiac Monitor, Model 1500 (CM-1500)
Brief Title: Evaluation of Physiological Variables and Detection of Blood Loss in Healthy Adults With Different Subject Positioning by the CM-1500
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZMS-1500-Pa2023
Record Dates: First submitted 2023-07-26; First posted 2023-08-07 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Fluid Loss; Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Supine Donation Position (Experimental)
  Interventions: Device: Whole blood donation supine
- Reclined Donation Position (Experimental)
  Interventions: Device: Whole blood donation reclined

INTERVENTIONS:
Device: Whole blood donation supine — Subjects will undergo a 1-unit whole blood donation in a supine position
  Arms: Supine Donation Position
Device: Whole blood donation reclined — Subjects will undergo a 1-unit whole blood donation in a reclined position
  Arms: Reclined Donation Position

SUMMARY:
The study is a prospective, non-randomized, non-blinded, non-significant risk study enrolling up to 60 healthy adult subjects consented to undergo a 1-unit whole blood draw procedure. Subjects will wear the study device (CM-1500) while positioned in either a supine or reclined position during the blood draw and study-required physiological parameters will be captured pre-, during, and post-donation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Ability and willingness to comply with the study procedures and duration requirements
* 18 years of age or older
* Consented and eligible to undergo a single unit whole blood donation

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Undergone an amputation of any upper extremity
* Diagnosed with dextrocardia
* Subjects who have a pacemaker
* Subjects with body hair density which prevents adequate application of device electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Smith, MD; PhD, Principal Investigator — SunCoast Blood Centers
Locations (2):
- United States (2):
  - Vitalant Research Institute, Denver, Colorado
  - SunCoast Blood Centers, Bradenton, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supine Donation Position | Reclined Donation Position
Started | 60 | 60
Completed | 60 | 58
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Device Error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supine Donation Position | Reclined Donation Position | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (18.8) | 48.1 (18.3) | 50.2 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 31 | 35 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Impact of Subject Positioning on Percent Change of Heart Rate (HR) After Minor Blood Loss (e.g., 500mL)
Description: The objective of this study is to determine if manual blood loss of up to 500mL of blood affects heart rate. This will be measured by determining the percent change in HR before and after the Blood Draw. The percent change will be calculated separately for each Arm (reclined, supine). Based on previous studies, a positive outcome would be indicated by an increase in HR (i.e., positive percent change).
Time Frame: Recovery period following donation (10 minutes)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Supine Donation Position | Reclined Donation Position
Number analyzed (Participants) | 60 | 58
percent change | 10.7 (2.3) | 14.7 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the point of subject enrollment through a maximum of 24hrs following completion of participations (i.e., 48hrs).
Arm/Group | Supine Donation Position | Reclined Donation Position
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 1/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supine Donation Position (N=60) | Reclined Donation Position (N=60)
Yes - Procedure Related (General disorders) | 0 | 1 (1) — Subject became dizzy after post-procedure monitoring. Subject was provided juice and a salty snack and was fine upon discharge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT05980013/Prot_SAP_002.pdf